CLINICAL TRIAL: NCT00000351
Title: Cognitive Correlates of Substance Abuse, Part 2
Brief Title: Cognitive Correlates of Substance Abuse, Part 2 - 16
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Other Study IDs: NIDA-3-0010-16
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2002-12

CONDITIONS: Amphetamine-Related Disorders
MeSH Terms: conditions — Amphetamine-Related Disorders

SUMMARY:
Part II: Examine cognitive performance of stimulant abusers (methamphetamine and cocaine) during recovery by assessing their cognitive function at monthly intervals.

DETAILED DESCRIPTION:
Part II: Examine cognitive performance of stimulant abusers (methamphetamine and cocaine) during recovery by assessing their cognitive function at monthly intervals.

ELIGIBILITY:
Please contact site for information

Inclusion Criteria:

M/F. Meet DSM-IV criteria for stimulant dependence. Agree to conditions of the study and sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute